CLINICAL TRIAL: NCT05522543
Title: Comparison of Passive Translatoric Intervertebral Glides and Manual Segmental Traction in Patients With Mechanical Low Back Pain
Brief Title: Comparison of Passive Translatoric Intervertebral Glides and Manual Segmental Traction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01049 Mahnoor
Record Dates: First submitted 2022-08-04; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Mechanical Low Back Pain
Keywords: Mechanical Low Back Pain,Mobilizations.Traction
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment with manual segmental lumber traction (Experimental): Patient education (Postural correction, lifting, sitting and sleeping positions) • Hot Pack 10 mins
  • Manual lumbar Traction (L1-L5) for 15-20 sec x5 sets • Lumbar facet gapping (LFG) in side lying (10 sec 3 sets) and Lumbar rotational facet gapping (LRFG) in side lying (10 sec 3 sets) • .Core stability exercises (Knee to chest, bridges, prone press ups, cat and camel stretches) • Home plan
  Interventions: Other: Conventional treatment with Passive translatoric intervertebral glides
- Conventional treatment with passive translatoric intervertebral glides (Active Comparator): Patient education (Postural correction, lifting, sitting and sleeping positions) • Hot Pack 10 mins
  • PA Glides (Central and Transverse mobilizations) (10 sec each) x5 sets • Core stabilization exercise (Knee to chest, bridges, prone press ups, cat and camel stretches) • Home plan (bridges, knee to chest, cat and camel stretch and prone press ups
  Interventions: Other: Conventional treatment with manual segmental lumbar traction

INTERVENTIONS:
Other: Conventional treatment with Passive translatoric intervertebral glides — Patient education (Postural correction, lifting, sitting and sleeping positions) • Hot Pack 10 mins
  • PA Glides (Central and Transverse mobilizations) (10 sec each) x5 sets • Core stabilization exercise (Knee to chest, bridges, prone press ups, cat and camel stretches) • Home plan (bridges, knee to chest, cat and camel stretch and prone press ups
  Arms: Conventional treatment with manual segmental lumber traction
Other: Conventional treatment with manual segmental lumbar traction — Patient education (Postural correction, lifting, sitting and sleeping positions) • Hot Pack 10 mins
  • Manual lumbar Traction (L1-L5) for 15-20 sec x5 sets • Lumbar facet gapping (LFG) in side lying (10 sec 3 sets) and Lumbar rotational facet gapping (LRFG) in side lying (10 sec 3 sets) • .Core stability exercises (Knee to chest, bridges, prone press ups, cat and camel stretches) • Home plan
  Arms: Conventional treatment with passive translatoric intervertebral glides

SUMMARY:
The aim of this study is to find and compare the effects of passive translatoric intervertebral glides and manual segmental traction in patients with mechanical low back pain on pain ,range of motion and disability. Randomized controlled trial done at Aziz Bhatti Shaheed teaching hospital Gujrat. Total 34 participants will be enrolled (17 in each group A and group B. Group A received PA glides while group B received manual traction 25-65 years participants were included in study. Study duration was of 3 months .Sampling technique applied was purposive non probability sampling technique. Tools used in the study are (NPRS),Modified Oswestry disability index. Data was analyzed through SPSS 22.

DETAILED DESCRIPTION:
Low back pain is a global health issue and one of the leading causes of disability and morbidity worldwide. The overall lifetime prevalence of low back pain is estimated to be as high as 60%-84% .According to some studies low back pain is more common in women (60.9%)than in men (39.1%). In which 97% of the cases were reported to be of mechanical in origin. Mechanical back ache is the low back pain without any recognizable pathology. It can originate from spinal structures such as bone, joints, disc, and nervous or soft tissue. Mechanical back pain can be acute or chronic. Persistent pain for less than 4 to 6 weeks can be termed as acute mechanical low back pain or lumbago while pain lasting for more than 6 weeks is called chronic back pain. The episodes of disabling chronic low back pain has a tendency to reoccur and it affects up to 23% of the population globally with 24% to 84% of recurrence rate annually .

In a recent narrative article published by in 2020, current rehabilitation strategies available for low back pain were reviewed. Various approaches are patient advice, regular physical exercises, McKenzie method, lumbar stabilization exercises, directional preference exercises, Yoga, strength building and aerobic exercises, traditional Chinese practices including Tai-chi and Qigong exercises, spinal mobilization and manipulation, Traction, Hot and cold therapy, bracing and rest.

Joint mobilizations have been used for the treatment of musculoskeletal pain and to increase functionality for many years. The exact physiological mechanism by which intervertebral joint mobilizations reduce nociceptive activity in spinal lesion is still unknown but due to recent advancement in technology most of the researches believe it can be due to the stimulation of mechanoreceptors as well as free fluid movement within the joint space and disc structures .

In 1960s Maitland proposed a classification system for these joint mobilizations which is not only a treatment method but also a diagnostic tool that can be used to diagnose a joint dysfunction based on clinical findings.

A study in 2015 by Karina Yuko analyzed that use of Maitland's PA glides for 30 seconds in each painful lumbar vertebra twice a week for 4 weeks significantly increased strength and mobility and reduced pain after the 2nd week of intervention.

A study conducted in Pakistan by Komal et al in 2018 showed that Maitland's grade I and II spinal glides are effective in reducing pain in patients with chronic low backache and can be used as an effective treatment in low back pain management .

In 2018, a study published spinal mobilization and gliding techniques were found to be more effective in reducing pain than other active therapies including exercises (p<0.05) while these were not comparatively effective in reducing disability (p>0.05). When compared with manipulation technique, spinal manipulation was considered more effective than spinal mobilization and intervertebral glides in treating low back pain .

In 2017, conducted a systematic review with meta-analysis on lumbar stabilization exercises and conventional physical therapy along with manual therapeutic approaches for low back pain and concluded that no one form of exercise is more effective than the other in treating the pain or disability and encouraged using both forms of techniques in rehabilitation of musculoskeletal disorders .

While there are numerous treatment options available, one of the common practices used for treatment of low back pain is spinal traction. Spinal traction is a technique in which, depending on the mode of delivery, varying amount of force is used to separate the vertebrae. It provides pain relief by removing the pressure off the spinal structures as well as by neurophysiological effects such as pain modulation of nociceptive input. This is generally believed that traction benefits the patients with acute back pain with neurological deficits as well as spinal stiffness. Available evidences suggest that even a small dose of traction (5-10kg)or 10-20% of total body weight proves to be effective. While another study supports that the optimal force of traction should be 40% of the total body weight .Traction can be applied in various ways that include mechanical or motorized traction via pulley system, auto-traction without external help of the therapist, gravitational traction with a suspension device or a manual traction with force applied by therapist.

A cross sectional survey was conducted in 2015 to estimate the number of physical therapists who use traction in their clinical practices. 4000 physical therapists were randomly included in the study. The response rate was 25.5% from which 76.6% reported using traction. Most of those who used spinal traction in their practice preferred manual delivery methods (68.3%) while the others used mechanical traction tables along with other conventional physiotherapy interventions like posture correction or stabilizing exercises.

In 2020 a trial to report the immediate effects of lumbar traction in patients with chronic low back pain. A total 40% to 50% of the body weight for mechanical traction was used and the mode of delivery was intermittent traction with or without vibrations. The results showed that lumbar traction with the force of 40% of total body weight especially along with vibration can be an effective intervention in chronic low back pain.

As discussed earlier the causes of mechanical low back pain are vertebral joint degeneration, disc pathologies, spinal muscular imbalances or strains and nerve tissue irritation, therefore intervertebral translatoric glides and lumbar manual segmental traction can be effective for pain management and restricted joint mobility. While currently to our knowledge there exists very weak evidence to which one technique can proved to be more effective than the other. Therefore this study will evaluate the efficacy of both the interventions in pain, restricted range of motion and disability in patients with mechanical low back pain,

ELIGIBILITY:
Inclusion Criteria:

Gender: Both Men and Women

* Age: 25 to 65 years
* Patients with mechanical low back pain and restricted lumbar movements for more than 3 months
* No neurological deficits
* No muscle weakness less than 4/5 during manual muscle testin

Exclusion Criteria:

Pregnancy

* People with history of inflammatory MSK disorders like ankylosing spondylitis and Rheumatoid arthritis etc.
* Patient with neuromuscular disorders
* Other Musculoskeletal deformity
* Acute Trauma
* Malignancy
* Patients on medications for Cardiac failure
* Class III BMI

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Modified Oswestry disability Index( MODI) | Changes from the Baseline, at 2nd week and at 4th week.
  MODI is a measure of disability that is a Gold standard tool for measuring functional outcome in low back pain. It is also used to discriminate between broad categories of back pain patients and it is useful to measure treatment outcomes. It is divided into ten sections that assess the level of pain and interference with physical activities such as sleeping, standing, walking, home making, social life and traveling. Each question has a possible six responses which are scored from 0 to 5. Patients check one response statement in each section that is most relevant to them. The score for each section is added and divided by the total possible score (fifty if all sections are completed), with the resulting score multiplied by a hundred to yield a percentage score with 0% equivalent to no disability and 100% equivalent to a great deal of disability.

SECONDARY OUTCOMES:
NPRS 0 to 10 | Changes from the Baseline, at 2nd week and at 4th week.
  NPRS is the 11 point questionnaire that is used to assess the pain. The patient is instructed to choose a number from 0 to 10 that best describes their pain. 0 would mean "no pain" and 10 would mean "worst possible pain".
  * 1 to 4: Mild pain
  * 5 to 6: Moderate
  * 7 to 10: severe The final rating will be the average of the 3 ratings taken during the last 24 hours.

OTHER OUTCOMES:
The joint range of motion assessed by Goniometer | Changes from the Baseline, at 2nd week and at 4th week.
  The goniometer is a device used to measure joint range of motion. It comprises of a body with 2 arms attached to it. One is fixed and the other is movable. The measure of ROM is performed by direct reading of the angle between the axis of rotation at the end of active ROM of the movement being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PHD, Principal Investigator — Riphah International University
Locations (1):
- Aziz Bhatti Shaheed teaching Hospital, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No